CLINICAL TRIAL: NCT00739375
Title: The Effect of Blood Flow in the Maturing Arteriovenous Access for Hemodialysis on the Development of Pulmonary Hypertension.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Ilya Goldin, Dr, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 112
Record Dates: First submitted 2008-08-17; First posted 2008-08-21 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Pulmonary Hypertension
Keywords: Influence; of av access; flow; development
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Primary arterio-venous vascular access creation — Primary arterio-venous vascular access creation, ECHO with pulmonary artery pressure measurements, Assessment of blood NO metabolite levels

SUMMARY:
Pulmonary hypertension (PHT) is an elevation of pulmonary arterial pressure (PAP) that can be the result of heart, lung or systemic disease. PHT also complicates chronic hemodialysis (HD) therapy immediately after the creation of an arteriovenous (AV) access, even before starting HD therapy. It tends to regress after temporary AV access closure and after successful kidney transplantation. Affected patients have significantly higher cardiac output. This syndrome is associated with a statistically significant survival disadvantage. The laboratory hallmark of this syndrome is reduced basal and stimulatory nitric oxide (NO) levels. It appears that patients with end-stage renal disease (ESRD) acquire endothelial dysfunction that reduces the ability of their pulmonary vessels to accommodate the AV access-mediated elevated cardiac output, exacerbating the PHT. Doppler echocardiographic screening of ESRD patients scheduled for HD therapy for the occurrence of PH is indicated. Early diagnosis enables timely intervention, currently limited to changing dialysis modality such as peritoneal dialysis or referring for kidney transplantation.An echocardiographic diagnosis of pulmonary hypertension (PHT) is made when the systolic pulmonary arterial pressure (PAP) exceeds normal values (30 mmHg). In mild PHT, PAP values range up to 45 mmHg, in moderate PHT, PAP is between 45 and 65 mmHg, and in severe PHT, PAP values are greater than 65 mmHg. Systolic PAP equals cardiac output times pulmonary vascular resistance (PVR), (i.e., PAP = cardiac output × PVR). Increased cardiac output by itself does not cause PH because of the enormous capacity of the pulmonary circulation to accommodate the increase in blood flow. Therefore development of PHT requires pathologic, marked elevation of pulmonary vascular resistance. The presence of PH may reflect serious pulmonary vascular disease, which can be progressive and fatal. Consequently, an accurate diagnosis of the cause of PHT is essential in order to establish an effective treatment program. Pulmonary hypertension can occur from diverse etiologies. In 1996 we first noted unexplained PH in some long-term hemodialysis (HD) patients during an epidemiologic study of this disorder (Nakhoul F and Yigla M Rambam Medical Cemter-Haifa). It was assumed that their PHT was related to end-stage renal disease (ESRD) or to long-term HD therapy via an arteriovenous (AV) access.

There are several potential explanations for the development of PHT in patients with ESRD. Hormonal and metabolic derangement associated with ESRD might lead to vasoconstriction of pulmonary vessels and increased pulmonary vascular resistance. Values of PAP may be further increased by high cardiac output resulting from the AV access itself, worsened by commonly occurring anemia and fluid overload. Despite almost five decades of HD therapy via a surgically created, often large, hemodynamically significant AV access the long-term impact of this intervention on the pulmonary circulation has received little attention.

RD versus AV HD via AV access

Proposed Mechanisms:

1. Elevated Parathyroid hormone
2. Metastatic Calcification due to the increase of the calcium-phosphor multiple
3. High cardiac output
4. Nitric oxide-endothelin metabolism
5. A-v Access flow

These observations indicate a role for AV access-mediated elevations in cardiac output in the pathogenesis of PH. The correlation between access flow and PAP values has not yet been studied. Since patients undergoing HD therapy via AV access had PH that reversed after successful kidney transplantation and after short AV access compression, we concluded that both ESRD and AV access-mediated elevated cardiac output are required for the development PH. From a physiologic point of view, due to the enormous capacity of the pulmonary microcirculation, increased cardiac output by itself cannot cause PH. It is the inability of the pulmonary circulation of some ESRD patients to accommodate the AV access-mediated elevated cardiac output that leads to the development of PH.

ELIGIBILITY:
Inclusion Criteria:

* All new primary av access

Exclusion Criteria:

* Preoperatively known pulmonary hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Correlation between av access flow and development of pulmonary hypertension | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Goldin, Dr, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel